CLINICAL TRIAL: NCT05719467
Title: A Double-blind Randomized Placebo-controlled Four-arm Trial to Assess the Efficacy of Oral Bicarbonate and Intravenous Butylscopolamine Bromide to Facilitate Spontaneous (Non-operative) Delivery in Pregnant Female Participants With Induction of Labor
Brief Title: SAINT: Safe Induction of Labor Trial
Acronym: SAINT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trond Melbye Michelsen, Professor, Senior Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 235247
Record Dates: First submitted 2022-12-18; First posted 2023-02-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Labor Complication; Induced; Birth; Pregnancy Related
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Butylscopolammonium Bromide; Sodium Bicarbonate; Tablets; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Buscopan and bicarbonate (Active Comparator)
  Interventions: Drug: Buscopan 20 MG/ML Injectable Solution; Drug: Sodium bicarbonate
- Buscopan and placebo (Active Comparator)
  Interventions: Drug: Buscopan 20 MG/ML Injectable Solution; Drug: Placebo
- Placebo and bicarbonate (Active Comparator)
  Interventions: Drug: Sodium bicarbonate; Drug: Nacl 0.9%
- Placebo and placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Nacl 0.9%

INTERVENTIONS:
Drug: Buscopan 20 MG/ML Injectable Solution — 1 mL intravenously
  Arms: Buscopan and bicarbonate; Buscopan and placebo
Drug: Sodium bicarbonate — 4 g orally
  Arms: Buscopan and bicarbonate; Placebo and bicarbonate
Drug: Placebo — 4g orally
  Other Names: Oral Tab
  Arms: Buscopan and placebo; Placebo and placebo
Drug: Nacl 0.9% — 1 mL intravenously
  Other Names: Intravenous placebo
  Arms: Placebo and bicarbonate; Placebo and placebo

SUMMARY:
Over the past years, the rates of labor induction have increased steadily, and at present more than one in four births occurs after induced labor in Norway. There is evidence that several groups of women benefit from labor induction, including those with preeclampsia (1), postdate pregnancy, diabetes, a large-for-gestational-age fetus, gestational diabetes, prelabor rupture of membranes at term, preterm prelabor rupture of membranes, twin pregnancy and intrahepatic cholestasis of pregnancy.

At the same time, induction of labor is an independent risk factor for adverse obstetric outcomes, including cesarean section, operative vaginal delivery, chorioamnionitis, labor dystocia, prolonged labor, uterine rupture, and neonatal pH < 7.10. A recent Norwegian nationwide clinical practice pilot evaluation demonstrated that the rate of intervention was high, and that as many as 44% of women with labor induction experienced operative delivery.

Given that induction of labor is a common procedure (15 000 women per year in Norway) and increases risk of several major obstetric complications, interventions that may reduce operative births and facilitate safe deliveries are highly warranted.

Bicarbonate and butylscopolamine bromide have been used in smaller studies in order to shorten labor. The medications seem to be safe with a low frequency of adverse events.

The rationale of the present study is therefore to assess the efficacy of oral bicarbonate and intravenous butylscopolamine bromide on facilitating spontaneous (non-operative) delivery in pregnant female participants with induction of labor.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be between 18 and 50 years of age at the time of signing the informed consent.
2. Participants who are female, pregnant, nulliparous and at or above 37 weeks of gestation
3. Participants who fulfill hospital criteria for induction of labor, and where a decision to induce labor has been made
4. Participants carrying a fetus in vertex position
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria:

1. Multiple gestation
2. Elective cesarean section
3. Spontaneous start of labor
4. Known maternal intestinal stenosis, ileus or megacolon
5. Persisting maternal tachycardia (heart rate > 130 beats per minute) >30 minutes continuously.
6. Known maternal myasthenia gravis
7. Persisting fetal tachycardia (fetal heart rate baseline > 170 beats per minute) >30 minutes continuously.
8. Maternal hypersensitivity to any of the ingredients in IMP (butylscopolamine bromide, bicarbonate or sodium chloride)
9. Women with heart disease who are under surveillance with heart rate monitoring during labor
10. Known fetal heart disease or known fetal malformations in the gastrointestinal system
11. Untreated maternal glaucoma
12. Maternal electrolyte disturbance: severe hyponatremia, severe hypokalemia
13. Maternal moderate/severe kidney failure (stage III-V: glomerulus filtration rate <59 ml/minute/1.73m2 )
14. Maternal elevated serum creatinine (>90umol/L)
15. Maternal elevated Alanine Aminotransferase (ALAT) >100 U/L. Participation can still be considered for participants with ALAT >100 U/L if explained by obstetric cholestasis or HELLP syndrome.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Spontaneous vs operative birth | Through study completion, an average of one week
  Number of participants with operative birth as compared to spontaneous birth

CONTACTS AND LOCATIONS:
Overall Officials: Trond M Michelsen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (5):
- Norway (5):
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital Rikshospitalet, Oslo
  - Oslo University Hospital Ullevål, Oslo
  - Stavanger University Hospital, Stavanger
  - The University Hospital of North Norway, Tromsø

REFERENCES:
- [Derived] Sorbye IK, Gunnes N, Solhoff AV, Haavaldsen C, Kessler J, Kjollesdal AM, Jacobsen AF, Magnussen EB, Pettersen ATR, Sande RK, Sjoborg KD, Ween-Velken ME, Leeves LT, Michelsen TM; SAINT Consortium. Multicentre double-blind randomised placebo-controlled four-arm trial to assess the effect of oral sodium bicarbonate and intravenous hyoscine butylbromide on spontaneous delivery after induction of labour in nulliparous women: protocol for the Safe Induction of Labour Trial (SAINT). BMJ Open. 2025 Mar 3;15(3):e093992. doi: 10.1136/bmjopen-2024-093992. PMID 40032397